CLINICAL TRIAL: NCT02410512
Title: A Phase Ib, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of MOXR0916 and Atezolizumab in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Assess the Safety and Pharmacokinetics of MOXR0916 and Atezolizumab (Also Known as MPDL3280A or Anti-PD-L1) in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO29674; 2015-000516-18 (EudraCT Number)
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — atezolizumab; Antibodies

ARMS (2):
- Dose Escalation: MOXR0916 + Atezolizumab (Experimental): Cohorts of at least 3 participants each will be treated at escalating doses of MOXR0916 in combination with a fixed dose of atezolizumab to determine the MTD or maximum administered dose (MAD).
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 [PD-L1] antibody; Drug: MOXR0916, a humanized agonist anti-OX40 monoclonal antibody
- Expansion: MOXR0916 + Atezolizumab (Experimental): Approximately 250-580 participants will be enrolled in the expansion stage to better characterize the safety, tolerability, pharmacokinetic variability, biomarkers of anti-tumor activity, and preliminary efficacy of MOXR0916 + atezolizumab in different cancer types.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 [PD-L1] antibody; Drug: MOXR0916, a humanized agonist anti-OX40 monoclonal antibody

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 [PD-L1] antibody — Atezolizumab will be administered intravenously.
  Other Names: Tecentriq
Drug: MOXR0916, a humanized agonist anti-OX40 monoclonal antibody — MOXR0916 will be administered intravenously.

SUMMARY:
This Phase Ib, open-label, dose-escalation study will evaluate the safety, tolerability, and pharmacokinetics of the combination of MOXR0916 and atezolizumab in participants with locally advanced, recurrent, or metastatic incurable solid malignancy that has progressed after available standard therapy; or for which standard therapy has proven to be ineffective or intolerable or is considered inappropriate; or for which a clinical trial of an investigational agent is a recognized standard of care. Participants will be enrolled in two stages: a dose-escalation stage and an expansion stage.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy of at least 12 weeks
* Adequate hematologic and end organ function
* Histologic documentation of locally advanced, recurrent, or metastatic incurable solid malignancy that has progressed after available standard therapy; or for which standard therapy is ineffective, intolerable, or considered inappropriate; or for which a clinical trial of an investigational agent is recognized standard of care
* Tumor specimen availability
* Measurable disease according to RECIST v1.1

Exclusion Criteria:

* Any anti-cancer therapy, whether investigational or approved, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks prior to initiation of study treatment
* Malignancies other than disease under study within 5 years prior to D1 of C1
* Primary central nervous system (CNS) malignancy, or untreated/active CNS metastases
* History of leptomeningeal disease
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug-induced), organizing pneumonia, or evidence of active pneumonitis on screening chest computed tomography scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* History of autoimmune disease
* Positive human immunodeficiency virus test result
* Active hepatitis B, hepatitis C, or tuberculosis
* Severe infection within 4 weeks prior to D1 of C1
* Prior allogeneic bone marrow or solid organ transplantation
* Significant cardiovascular disease
* Known clinically significant liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2015-04-24 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose-Limiting Toxicities (DLTs) | Days (D) 1-21 of Cycle (C) 1 (cycle = 21 days); up to D42 if extended monitoring warranted
Number of Participants with Adverse Events Graded per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 4.0 | Baseline until 90 days after last dose or initiation of another systemic anti-cancer therapy, whichever occurs first (up to 3 years)

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) of MOXR0916 | Up to 1 year
Recommended Phase II Dose (RP2D) of MOXR0916 | Up to 1 year
Percentage of Participants with Anti-MOXR0916 and Anti-Atezolizumab Antibodies | Up to 120 days after the treatment discontinuation visit
Number of Cycles Received with MOXR0916 | Baseline until treatment discontinuation (up to 3 years)
Dose Intensity of MOXR0916 | Baseline until treatment discontinuation (up to 3 years)
Area under the Concentration-Time Curve (AUC) of MOXR0916 | Up to 120 days after the treatment discontinuation visit
Serum Maximum Observed Concentration (Cmax) of MOXR0916 | Up to 120 days after the treatment discontinuation visit
Serum Minimum Observed Concentration (Cmin) of MOXR0916 | Up to 120 days after the treatment discontinuation visit
Clearance (CL) of MOXR0916 | Up to 120 days after the treatment discontinuation visit
Volume of Distribution at Steady State (Vss) of MOXR0916 | Up to 120 days after the treatment discontinuation visit
Serum Cmax of Atezolizumab | Up to 120 days after the treatment discontinuation visit
Serum Cmin of Atezolizumab | Up to 120 days after the treatment discontinuation visit
Percentage of Participants with Objective Response Determined Using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Baseline until disease progression (up to 3 years)
Duration of Objective Response (DOR) Determined Using RECIST v1.1 | From first objective response until death or relapse per RECIST v1.1, whichever occurs first (up to 3 years)
Progression-Free Survival (PFS) Determined Using RECIST v1.1 | Baseline until death or disease progression per RECIST v1.1, whichever occurs first (up to 3 years)
Percentage of Participants with Objective Response Determined Using Modified RECIST | Baseline until disease progression (up to 3 years)
DOR Determined Using Modified RECIST | From first objective response until death or relapse per RECIST v1.1, whichever occurs first (up to 3 years)
PFS Determined Using Modified RECIST | Baseline until death or disease progression per RECIST v1.1, whichever occurs first (up to 3 years)
Overall Survival (OS) | Baseline until death (up to 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- United States (9):
  - HonorHealth Research Institute - Bisgrove, Scottsdale, Arizona
  - University of Colorado, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - University Of Chicago Medical Center; Section Of Hematology/Oncology, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Can Ins, Boston, Massachusetts
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Austin Hospital, Heidelberg, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (3):
  - Institut Jules Bordet, Anderlecht
  - UZ Gent, Ghent
  - Sint Augustinus Wilrijk, Wilrijk
- Canada (3):
  - British Columbia Cancer Agency (Bcca) - Vancouver Cancer Centre, Vancouver, British Columbia
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
- Gustave Roussy, Villejuif, France
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Yonsei University Health System/Severance Hospital, Seoul
- Spain (4):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hosp de Madrid Norte Sanchinarro; Centro Integral; Onco Clara Campal, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia